CLINICAL TRIAL: NCT05214378
Title: High Frequency Sacral Root Stimulation to Improve Bladder and Bowel Emptying Following SCI
Brief Title: High Frequency SARS for Neurogenic Bladder and Bowel Emptying
Acronym: SARS600
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B4085-P
Record Dates: First submitted 2022-01-21; First posted 2022-01-28 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Testing alternative stimulation patter in a set of individuals who are already implanted with device. Study participants will act as their own controls comparing outcomes with and without the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Arm (Experimental): The investigators will test an alternative pattern of sacral root stimulation in individuals who are already implanted with the device. Study participants will act as their own controls.
  Interventions: Device: Finetech-Brindley Sacral Anterior Roots Stimulation System

INTERVENTIONS:
Device: Finetech-Brindley Sacral Anterior Roots Stimulation System — Electrodes implanted on sacral roots connected to implanted induction coil. External controller box administers stimulation via induction through skin to electrodes. Stimulation activates nerves to modulate bladder, bowel, and sexual functions.
  Other Names: Vocare

SUMMARY:
The purpose of this study is to determine if bladder emptying can be achieved using stimulation of the sacral roots at certain frequencies. Neurogenic bladder dysfunction occurs after spinal cord injury (SCI). It is a problem that often includes detrusor-sphincter-dyssynergia (DSD), which results in difficulty emptying the bladder due to reflex urethral sphincter contractions during bladder emptying. Individuals with DSD typically require a catheter to empty their bladder. Some people have received an implanted device that stimulates the spinal nerves that connect to the bladder to empty the bladder without a catheter. However, this procedure usually also includes cutting nerves to stop unwanted reflexes. For this study, the investigators are testing a new stimulation pattern to determine if it can help achieve bladder emptying without having to cut nerves. Individuals with SCI who have received an implanted sacral root stimulation device are being asked to participate in this research to test the effectiveness of electrical stimulation to relax the urethral sphincter and promote bladder emptying.

DETAILED DESCRIPTION:
Background: Spinal cord injury (SCI) leads to neurogenic bladder dysfunctions, and often includes difficulty with emptying the bladder due to detrusor-sphincter dyssynergia (DSD). Current bladder management strategies include catheterization, pharmaceuticals, and/or surgery, but these interventions insufficiently meet individuals' needs. The neurogenic bladder can be emptied using sacral anterior root stimulation (SARS) with electrodes implanted on the sacral nerves to produce bladder contractions. However, this emptying can be impeded by reflex contractions of the urethral sphincter. The sacral sensory roots are typically transected (rhizotomy) to reduce these reflex contractions, but this rhizotomy also impairs desirable reflexes (e.g. sexual function) and sacral sensation if present. Experiments in animals have shown that sacral root stimulation at 600 Hz can inhibit urethral sphincter activity, which has the potential. This approach could be used in lieu of the rhizotomy to improve bladder emptying efficiency.

Objective: The objective of this study is to test the feasibility and potential effectiveness of 600 Hz sacral root stimulation to limit urethral sphincter activity in individuals with neurogenic bladder dysfunction. The investigators hypothesize that sacral root stimulation at 600 Hz will result in lower urethral sphincter pressures compared to pressures in response to stimulation at the lower frequencies that are typically used for SARS.

Study Design: In this feasibility study, the investigators will enroll 8 participants, male or female, who have SCI and who already use implanted sacral root anterior stimulation to manage their bladder. Participants will act as their own controls. Stimulus waveforms for urethral sphincter inhibition will be tested in the clinical laboratory in a single session. The investigators will not need to conduct new surgeries or implant procedures. The primary outcome measure is urethral sphincter pressure, and additional outcome measures include bladder pressure, rectal pressure, and bladder volume as measured in clinically standard urodynamics examination.

Clinical Impact: This approach could help restore bladder function by reducing urethral sphincter activity that impedes bladder emptying for individuals with SCI. The investigators could improve approaches for promoting bladder emptying by eliminating the need for sacral posterior rhizotomy.

ELIGIBILITY:
Inclusion Criteria:

* Uses a SARS System for bladder management
* Suprasacral SCI
* Neurologically stable
* Skeletally mature

Exclusion Criteria:

* Active sepsis
* Open pressure sores on or around pelvis
* Bleeding diathesis
* Significant urethral trauma, erosion, or stricture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Bourbeau, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (2):
- United States (2):
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Urethral Sphincter Pressure
Description: urethral sphincter pressure measured in response to presence of stimulation (treatment) compared to pressure in absence of stimulation
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Treatment Arm
Number analyzed (Participants) | 4
cmH2O | 50 (45)

ADVERSE EVENTS:
Time Frame: 1 week
Description: Procedures performed included clinical standard urodynamics, which is a diagnostic exam, and mild electrical stimulation using a device that the participant already used for their bladder management. Participants were not considered at risk of mortality associated with this study.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT05214378/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT05214378/ICF_000.pdf